CLINICAL TRIAL: NCT04995588
Title: Role of Innate T Cells in Physiopathology of Systemic Sclerosis
Brief Title: Systemic Sclerosis and Innate T Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Sclero-LTI
Record Dates: First submitted 2021-07-23; First posted 2021-08-09 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2023-09

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood test (Other): Unique blood test for all the participants included in the study to constitute a local biobank to assess in a grouped manner the prespecified outcomes
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — Unique blood draw of 45mL for all the participants

SUMMARY:
Innate T cells (ITC) are decreased in systemic sclerosis (SS) and an early lymphocyte innateness has been reported. In the other part, ITC are implicated on inflammatory process, including the IL-33/ST2 axis, which is also involved in ScS endotheliopathy.

Data are however scarce and physiopathological mechanisms have not been assessed to date.

The investigators hypothesize a global lymphocyte innateness in SSc, linked to a chronic ITC stimulation by innate signals leading to ITC exhaustion, and their potential role in endotheliopathy and fibroblast activation in SSc.

ELIGIBILITY:
Inclusion Criteria:

* SSc according to the 2013 ACR/EULAR 2013 criteria (or the 2001 Leroy's criteria for early SSc)
* Patients with others connective tissue disease:

  * Systemic erythematosus lupus (SLE) according to the 2019 ACR/EULAR criteria
  * Primary Sjögren syndrome (pSS) according to the 2016 ACR/EULAR criteria
  * Rheumatoid arthritis according to the 2010 ACR/EULAR criteria
  * Idiopathic inflammatory myopathy (IIM) according to the 2017 ACR/EULAR criteria
* Healthy subjects from general population without known autoimmune disease or connective tissue disease
* ≥18 years-old

Exclusion Criteria:

* Overlap syndrome (including secondary Sjögren syndrome)
* Weight <55 kgs
* Known primary cell immunodeficiency
* Past of autologous or allogenic hematopoietic stem cell transplantation
* Solid neoplasia or malignant hemopathy in remission for less than 12 months an
* Chemotherapy and/or immune checkpoint inhibitors in the last 12 months
* Systemic retinoids
* Active infection and/or antibiotics in the last 2 weeks
* Known active chronic infection among HIV, HTLV, viral hepatitis, syphilis
* Vaccination in the last 4 weeks
* Subject refusing genetic analysis for the present study
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2025-08-28 (Estimated); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
Basal numeration of circulating ITC (iNKT, MAIT, γδ-T and innate CD8(+) T-cells) | Through study completion, an average of 1 year
  Percentage AND absolute count of iNKT, MAIT, γδ-T and innate CD8(+) T- cells in flow cytometry among total T cells in SSc patients (n=60), patients with other connective tissue disease (systemic lupus erythematosus, rheumatoid arthritis, primary Sjögren's syndrome, idiopathic inflammatory myopathies) (n=60), and in healthy subjects (n=60)
Basal expression level of Ki67 among circulating ITC (iNKT, MAIT, γδ-T and innate CD8(+) T-cells) | Through study completion, an average of 1 year
  Percentage of iNKT, MAIT, γδ-T and innate CD8(+) T-cells expressing Ki67 in flow cytometry in SSc patients (n=60), patients with other connective tissue disease (systemic lupus erythematosus, rheumatoid arthritis, primary Sjögren's syndrome, idiopathic inflammatory myopathies) (n=60), and in healthy subjects (n=60)
Basal expression level of PLZF AND Eomes AND T-bet AND Helios of circulating ITC (iNKT, MAIT, γδ-T and innate CD8(+) T-cells) | Through study completion, an average of 1 year
  Percentage of iNKT, MAIT, γδ-T and innate CD8(+) T-cells expressing PLZF, Eomes, T-bet and Helios in flow cytometry in SSc patients (n=60), patients with other connective tissue disease (systemic lupus erythematosus, rheumatoid arthritis, primary Sjögren's syndrome, idiopathic inflammatory myopathies) (n=60), and in healthy subjects (n=60)
Basal expression of perforin AND granzyme A among circulating ITC (iNKT, MAIT, γδ-T and innate CD8(+) T-cells) | Through study completion, an average of 1 year
  Percentage of iNKT, MAIT, γδ-T and innate CD8(+) T-cells expressing perforin and granzyme A in flow cytometry in SSc patients (n=60), patients with other connective tissue disease (systemic lupus erythematosus, rheumatoid arthritis, primary Sjögren's syndrome, idiopathic inflammatory myopathies) (n=60), and in healthy subjects (n=60)
IFN-ɣ, IL-4 and IL-17 production of iNKT, MAIT, γδ-T and innate CD8(+) T-cells in response to IL-1, IL-8, IL-12, IL-18, IL-33 and fractalkine | Through study completion, an average of 1 year
  Percentage of iNKT, MAIT, γδ-T and innate CD8(+) T-cells expressing IFN-ɣ AND IL-4 AND IL-17 in flow cytometry upon stimulation by various combinations of IL-1, IL-8, IL-12, IL-18, IL-33 and fractalkine in SSc patients (n=60), patients with other connective tissue disease (systemic lupus erythematosus, rheumatoid arthritis, primary Sjögren's syndrome, idiopathic inflammatory myopathies) (n=60), and in healthy subjects (n=60)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU poitiers, Poitiers, France